CLINICAL TRIAL: NCT06148506
Title: A Prospective NIS to Evaluate the Clinical Outcomes of Risarg® (Ribociclib) Combined With Endocrine Therapy or Chemotherapy in Patients With HR+HER2 - Advanced Breast Cancer in Routine Clinical Practice in the Russian Federation
Brief Title: A Prospective NIS to Evaluate the Clinical Outcomes of Risarg® (Ribociclib) Combined With Endocrine Therapy or Chemotherapy in Patients With HR+HER2 - aBC in Routine Clinical Practice in the Russia
Acronym: ValerEE
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011ARU04
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: HR+HER2- Advanced Breast Cancer
Keywords: HR+HER2- advanced breast cancer,; ribociclib+ET,; Chemotherapy; ribociclib; NIS
MeSH Terms: interventions — ribociclib; Drug Therapy, Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Ribociclib Arm: ribociclib (600 mg, 3 weeks on/1 week off)+ IA/FUL + goserilin for premenopausal patients
  Interventions: Other: Ribociclib
- Combination chemotherapy: The choice of which chemotherapy combination used on study is decided by the physician
  Interventions: Other: Combination chemotherapy

INTERVENTIONS:
Other: Ribociclib — There is no treatment allocation. Participants with HR+HER2- aBC that initiated treatment with ribociclib+ET by prescription within the study enrollment timeline will be recruited.
  Other Names: Risarg
  Groups: Ribociclib Arm
Other: Combination chemotherapy — There is no treatment allocation. Participants with HR+HER2- aBC that initiated treatment with CT by prescription within the study enrollment timeline will be recruited.
  Groups: Combination chemotherapy

SUMMARY:
This is а prospective, non-interventional, primary data collection cohort study to evaluate the clinical outcomes of the combination of ribociclib + ET and combination chemotherapy in the real-life setting in Russia. This study is observational in nature; it does not impose a therapy, diagnostic/therapeutic interventions or a visit schedule.

DETAILED DESCRIPTION:
Patients with HR+HER2- advanced breast cancer that initiated treatment with ribociclib+ET or combination CT will be enrolled. Approximately, 188 patients will be included into each treatment cohort of the study across different study sites in the Russian Federation and will be assigned to one of the below treatment arms:

* Ribociclib arm: ribociclib (600 mg, 3 weeks on/1 week off)+ IA/FUL + goserilin for premenopausal patients (N = 188)
* Combination chemotherapy arm: physician's choice (N = 188) The study will consist of pre-index period, index date and follow up period. Retrospective data will be collected as such: Medical history, previous treatment for Breast cancer (neoad'uvant and ad'uvant if applicable).In this study an index date is defined as a start of ribociclib+ET or chemotherapy treatment. Post-index follow-up period is 24 months or Progressive disease.

Patients will attend the sites in accordance with routine clinical practice. It is assumed according to the clinical practice that visits will be conducted every 3-4 months. Patients will undergo standard procedures and tests according to clinical guidelines and physician's judgement. No additional diagnostic or monitoring procedures will be applied to the patients and epidemiological methods shall be used for the analysis of collected data. Available data from routine clinical management of the patients will be collected at patients' visits to the clinical site. Patients enrolled in the study will be followed up until death or study close whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the moment of ribociclib+ET or CT initiation.
2. Female/Male gender.
3. Luminal A, Luminal B subtype.
4. Patients with ECOG performance status ≤ 2.
5. Confirmed diagnosis of locally advanced/metastatic not eligible to surgery HR+HER2- BC (de novo) for whom the treating physician took the decision to initiate treatment with ribociclib+IA/FUL or combination chemotherapy before entering the study in the first line of the treatment.
6. Multiple visceral metastases (including stable CNS mts).
7. Pre-/Pere /postmenopause.
8. Patient who initiated treatment with ribociclib+IA/FUL or combination chemotherapy no longer than 4 weeks (28 days) prior to written informed consent for this study.

Exclusion Criteria:

1. Patients with a life expectancy of less than 3 months per the investigator's judgment.
2. Patients participating in any interventional clinical trial that includes investigational or marketed products at the time of enrollment. (Patients participating in other investigator initiated research or NIS can be included as long as their standard of care is not altered by the study).
3. Patients on active treatment for malignancies other than aBC at the time of enrollment.
4. Patients who are unable to understand the nature of the study and are unwilling to sign an informed consent.
5. Patients with visceral crisis (according to ABC5 definition*) *Visceral crisis is defined as severe organ dysfunction, as assessed by signs and symptoms, laboratory studies and rapid progression of disease. Visceral crisis is not the mere presence of visceral metastases but implies important organ compromise leading to a clinical indication for the most rapidly efficacious therapy [8].

Examples: Liver visceral crisis: rapidly increasing bilirubin >1.5 ULN in the absence of Gilbert's syndrome or biliary tract obstruction. Lung visceral crisis: rapidly increasing dyspnoea at rest, not alleviated by drainage of pleural effusion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HR+HER2- advanced breast cancer that initiated treatment with ribociclib+ET or combination CT will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
time to treatment failure (TTF) | Up to 24 months
  The primary efficacy endpoint of the study is time to treatment failure (TTF) in in RIB + ET (AI/FUL) and combination chemotherapy cohorts. Time to treatment failure (TTF) is defined as the time from initiation of treatment to discontinuation of treatment for any reason, including disease progression, treatment toxicity, and death.

SECONDARY OUTCOMES:
Number of participants by menopausal status | Baseline
  Number of participants premenopausal, perimenopausal ad postmenopausal at baseline.
Number of participants by HER2 status | Baseline
  Number of participants by HER2 status (HER2 receptor positive/negative)
Number of participants by tumor, nodes and metastasis (TNM) stage | Baseline
  Number of participants by tumor, nodes and metastasis (TNM) stage
Chemotherapy regimens | Up to 24 months
  Percentage of patients receiving different combination chemotherapy regimens.
Time to treatment failure (TTF) in the subgroups | Dec2027
  Time to treatment failure in HR+HER2- aBC patients in RIB+ET and combination chemotherapy cohorts (in the subgroups Disease-free interval (DFI) ≤ 12 month, DFI > 12 month, Pre- and post menopause).
  Disease-free interval (DFI) will be calculated as the time from the date of diagnosis until the date of first recurrence/progression.
Objective response rate (ORR) | Up to 24 months
  Objective response rate (ORR) as assessed by the investigator. Objective response rate (ORR) is the proportion of patients with a best overall response of Complete Response or Partial Response.
Clinical benefit rate (CBR) | Up to 24 months
  Clinical benefit rate (CBR) as assessed by the investigator. Clinical benefit rate (CBR) is the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR) , or an overall lesion response of Stable Disease or Non-CR/Non-PD which lasts for a minimum time duration (with a default of at least 24 weeks in breast cancer studies).
Time to onset of response (TTR) | Up to 24 months
  Time to onset of response (TTR) as assessed by the investigator. Time to onset of response (TTR) is defined as the time from the date of randomization to the first documented response of either CR or PR, which must be subsequently confirmed (although date of initial response is used, not date of confirmation). CR and PR are based on tumor response data as per local review.
Assessment of Quality of life - EQ-5D-5L | Up to 24 months
  Quality of life (EQ-5D-5L) during treatment with ribociclib + ET (AI/FUL) and combination chemotherapy is measured, if used in real practice.
  The scale measures quality of life on a 5-component scale: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Russia (18):
  - Novartis Investigative Site, Kaluga, Russia
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nal'chik
  - Novartis Investigative Site, Podolsk
  - Novartis Investigative Site, Saransk
  - Novartis Investigative Site, Tambov
  - Novartis Investigative Site, Tver'
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Vladikavkaz
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No